CLINICAL TRIAL: NCT00992277
Title: In-vivo Analysis and Clinical Evaluation of the Performance of a Fractional CO2 Laser System (eMatrixCO2) Intended for Treatment of Soft Tissue
Brief Title: In-vivo Analysis and Clinical Evaluation of the Performance of a Fractional CO2 Laser System (eMatrixCO2)
Acronym: eMatrixCO2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DC75061
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Aesthetic Dermatology

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Facial (Experimental): Skin rejuvenation treatments
  Interventions: Procedure: Ablation and skin resurfacing

INTERVENTIONS:
Procedure: Ablation and skin resurfacing

SUMMARY:
This study will:

Evaluate the in vivo histological and molecular effects of treatment with eMatrixCO2 and to determine the dynamics of their development over time following treatment.

Determine the safety and efficacy of treatment with eMatrixCO2 for use in Aesthetic dermatological procedures requiring the ablation, vaporization, excision, incision, or coagulation of soft tissue.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent agreement signed by the subject.
* Healthy males or females older than 21 years of age.
* Fitzpatrick skin type I-V (Although the systems are cleared for all skin types I-VI, it is recommended to use the Matrix applicators on skin types I - V).
* Willingness to follow the treatment and follow-up schedule and the post-treatment care.
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* Pregnant and/or breastfeeding.
* Having a permanent implant in the facial skin area, such as an injected chemical substance - Not relevant for the abdominoplasty group.
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session.
* Use of retinoids, antioxidants or therapeutic skin nourishing supplements within 2 months of treatment or during the study and oral retinoids within 6 months of the study.
* Having received a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study- Not relevant for the abdominoplasty group.
* Having received treatment with light, RF or other devices in the treated area within 6 months of treatment or during the study.
* Having received Botox/collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 9 months of treatment or during the study.
* Having undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study- Not relevant for the abdominoplasty group.
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study.
* History of keloid scarring or of abnormal wound healing.
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: active acne, excessive skin dryness, psoriasis, eczema, rash, rosacea (particularly severe open wound stage), varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Suffering from hormonal imbalance, as per the Investigator's discretion.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including actinic keratosis, presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
* Vascular lesion, tattoo or permanent make-up in the treated area.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Participation in a study of another device or drug within three month prior to enrollment or during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Histological and molecular assessment of tissue taken following treatment with different parameters and at various time points | over time following treatment.
Record number and type of any AE during the study | study duration

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scripps Health, San Diego, California
  - South Dermatology Institute, Tustin, California
  - Zel Skin & Laser Specialists, Saint Edina, Minnesota